CLINICAL TRIAL: NCT05512000
Title: Increasing Word Learning Efficiency in Children Who Are Deaf and Hard of Hearing Through Retrieval Practice
Brief Title: Retrieval Practice for Word Learning for Deaf and Hard of Hearing Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jena McDaniel, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221204
Record Dates: First submitted 2022-08-11; First posted 2022-08-23 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Hearing Loss; Language Impairment
MeSH Terms: conditions — Hearing Loss; Language Disorders

STUDY DESIGN:
Intervention Model Description: Adapted alternating treatments research design with 3 conditions per participant. Four participants are randomly assigned to each contrast (arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Contrast A (Experimental): Feedback vs no feedback with massed trials
  Interventions: Behavioral: Feedback with massed trials; Behavioral: No feedback with massed trials; Behavioral: No teaching control
- Contrast B (Experimental): Feedback vs no feedback with spaced trials
  Interventions: Behavioral: Feedback with spaced trials; Behavioral: No feedback with spaced trials; Behavioral: No teaching control
- Contrast C (Experimental): Spaced vs massed trials without feedback
  Interventions: Behavioral: No feedback with massed trials; Behavioral: No feedback with spaced trials; Behavioral: No teaching control
- Contrast D (Experimental): Spaced vs massed trials with feedback
  Interventions: Behavioral: Feedback with massed trials; Behavioral: Feedback with spaced trials; Behavioral: No teaching control

INTERVENTIONS:
Behavioral: Feedback with massed trials — The participant receives feedback on their accuracy completing retrieval practice tasks. Exposures for one word are provided before moving to the next word in each session.
  Arms: Contrast A; Contrast D
Behavioral: Feedback with spaced trials — The participant receives feedback on their accuracy completing retrieval practice tasks. Exposures for each word are interspersed with one another (e.g., an exposure for word 1, then one for word 3, then one for word 2, etc.) in each session.
  Arms: Contrast B; Contrast D
Behavioral: No feedback with massed trials — The participant does not receive feedback on their accuracy completing retrieval practice tasks. Exposures for one word are provided before moving to the next word in each session.
  Arms: Contrast A; Contrast C
Behavioral: No feedback with spaced trials — The participant does not receive feedback on their accuracy completing retrieval practice tasks. Exposures for each word are interspersed with one another (e.g., an exposure for word 1, then one for word 3, then one for word 2, etc.) in each session.
  Arms: Contrast B; Contrast C
Behavioral: No teaching control — The words in this set are not taught, only assessed.

SUMMARY:
This study is designed to advance the promising yet underutilized research on retrieval practice by evaluating the effectiveness and efficiency of two key retrieval practice features (feedback and spacing). The study uses four single case adapted alternating treatments studies, each with four 5- to 8-year-old children who are deaf and hard of hearing to evaluate the effects of feedback and spacing on the efficiency of word learning and retention.

DETAILED DESCRIPTION:
The proposed research addresses a long-standing and important challenge of improving language skills of children who are deaf and hard of hearing, a historically under researched group. The study aims to leverage retrieval practice - an empirically validated intervention approach - for improving how efficiently children who are deaf and hard of hearing learn and retain new words. To advance the promising yet underutilized research on retrieval practice, the study completes the next logical step of evaluating the effectiveness and efficiency of two key retrieval practice features: feedback and spacing. Feedback is predicted to result in more efficient learning because it focuses attention on unmastered material, prevents the illusion of success, and reduces repeated errors. Spacing trials are predicted to result in more efficient learning than massed trials because they require more effort with fewer cues provided. The study will accomplish these aims through four single case adapted alternating treatments design studies with sixteen 5- to 8- year-old children who are deaf and hard of hearing. Study innovations include the critical evaluation of retention and use of a multi-session intervention context. The knowledge gained will guide language intervention for children who are deaf and hard of hearing.

ELIGIBILITY:
Inclusion Criteria:

* At least minimal prelingual hearing loss
* Standard scores of at least 70 for receptive and expressive vocabulary skills
* English is only spoken language

Exclusion Criteria:

* Below average nonverbal cognition
* Uncorrected vision impairment
* Evidence of severe motor impairment

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2023-02-05 (Actual); Primary Completion 2025-07-11 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Labeling - acquisition | End of intervention. The intervention ends when the participant achieves >75% accuracy 3 sessions in a row (up to 6 months).
  Percent accuracy labeling target words expressively (number of target words correctly labeled when shown the object divided by the number of words in the set [i.e., 4] times 100)
Labeling - retention | Four weeks after the intervention ends
  Percent accuracy labeling target words expressively (number of target words correctly labeled when shown the object divided by the number of words in the set [i.e., 4] times 100)

SECONDARY OUTCOMES:
Identifying - acquisition | End of intervention. The intervention ends when the participant achieves >75% accuracy for labeling 3 sessions in a row (up to 6 months).
  Percent accuracy identifying target words receptively (number of objects correctly identified when target word is named divided by the number of words in the set [i.e., 4] times 100)
Semantic - acquisition | End of intervention. The intervention ends when the participant achieves >75% accuracy for labeling 3 sessions in a row (up to 6 months).
  Percent accuracy labeling associated semantic information (i.e., location; number of target objects' locations correctly named when shown the object divided by the number of words in the set [i.e., 4] times 100)
Identifying - retention | Four weeks after the intervention ends
  Percent accuracy identifying target words receptively (number of objects correctly identified when target word is named divided by the number of words in the set [i.e., 4] times 100)
Semantic - retention | Four weeks after the intervention ends
  Percent accuracy labeling associated semantic information (i.e., location; number of target objects' locations correctly named when shown the object divided by the number of words in the set [i.e., 4] times 100)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Graphs with individual data points will be reported in manuscripts that share the primary study findings. Sharing of such graphical data will permit inclusion of the project's results in future meta-analyses.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available when manuscripts are published.
Access Criteria: Data will become available through the published manuscript(s).

REFERENCES:
- [Background] Antia SD, Lederberg AR, Easterbrooks S, Schick B, Branum-Martin L, Connor CM, Webb MY. Language and Reading Progress of Young Deaf and Hard-of-Hearing Children. J Deaf Stud Deaf Educ. 2020 May 30;25(3):334-350. doi: 10.1093/deafed/enz050. PMID 32052022
- [Background] Bjork, E. L., & Bjork, R. A. (2011). Making things hard on yourself, but in a good way: Creating desirable difficulties to enhance learning. Psychology and the Real World: Essays Illustrating Fundamental Contributions to Society, 2, 59-68.
- [Background] Bjork, R. A. (1994). Memory and metamemory considerations in the. Metacognition: Knowing About Knowing, 185.
- [Background] Bobzien, J. L., Richels, C., Schwartz, K., Raver, S. A., Hester, P., & Morin, L. (2015). Using repeated reading and explicit instruction to teach vocabulary to preschoolers with hearing loss. Infants & Young Children, 28(3), 262-280.
- [Background] Boons T, De Raeve L, Langereis M, Peeraer L, Wouters J, van Wieringen A. Expressive vocabulary, morphology, syntax and narrative skills in profoundly deaf children after early cochlear implantation. Res Dev Disabil. 2013 Jun;34(6):2008-22. doi: 10.1016/j.ridd.2013.03.003. Epub 2013 Apr 11. PMID 23584181
- [Background] Brennan-Jones CG, White J, Rush RW, Law J. Auditory-verbal therapy for promoting spoken language development in children with permanent hearing impairments. Cochrane Database Syst Rev. 2014 Mar 12;2014(3):CD010100. doi: 10.1002/14651858.CD010100.pub2. PMID 24619508
- [Background] Carpenter SK. Cue strength as a moderator of the testing effect: the benefits of elaborative retrieval. J Exp Psychol Learn Mem Cogn. 2009 Nov;35(6):1563-9. doi: 10.1037/a0017021. PMID 19857026
- [Background] Carpenter, S. K., & Yeung, K. L. (2017). The role of mediator strength in learning from retrieval. Journal of Memory and Language, 92, 128-141.
- [Background] Coyne JH, Borg JM, DeLuca J, Glass L, Sumowski JF. Retrieval practice as an effective memory strategy in children and adolescents with traumatic brain injury. Arch Phys Med Rehabil. 2015 Apr;96(4):742-5. doi: 10.1016/j.apmr.2014.09.022. Epub 2014 Oct 13. PMID 25312580
- [Background] Fritz CO, Morris PE, Nolan D, Singleton J. Expanding retrieval practice: an effective aid to preschool children's learning. Q J Exp Psychol (Hove). 2007 Jul;60(7):991-1004. doi: 10.1080/17470210600823595. PMID 17616915
- [Background] Geers AE, Mitchell CM, Warner-Czyz A, Wang NY, Eisenberg LS; CDaCI Investigative Team. Early Sign Language Exposure and Cochlear Implantation Benefits. Pediatrics. 2017 Jul;140(1):e20163489. doi: 10.1542/peds.2016-3489. Epub 2017 Jun 12. PMID 28759398
- [Background] Geers AE, Sedey AL. Language and verbal reasoning skills in adolescents with 10 or more years of cochlear implant experience. Ear Hear. 2011 Feb;32(1 Suppl):39S-48S. doi: 10.1097/AUD.0b013e3181fa41dc. PMID 21832889
- [Background] Goossens, N. A., Camp, G., Verkoeijen, P. P., & Tabbers, H. K. (2014). The effect of retrieval practice in primary school vocabulary learning. Applied Cognitive Psychology, 28(1), 135-142.
- [Background] Haebig E, Leonard LB, Deevy P, Karpicke J, Christ SL, Usler E, Kueser JB, Souto S, Krok W, Weber C. Retrieval-Based Word Learning in Young Typically Developing Children and Children With Development Language Disorder II: A Comparison of Retrieval Schedules. J Speech Lang Hear Res. 2019 Apr 15;62(4):944-964. doi: 10.1044/2018_JSLHR-L-18-0071. PMID 30986145
- [Background] Jones, A. C., Wardlow, L., Pan, S. C., Zepeda, C., Heyman, G. D., Dunlosky, J., & Rickard, T. C. (2016). Beyond the rainbow: Retrieval practice leads to better spelling than does rainbow writing. Educational Psychology Review, 28(2), 385-400.
- [Background] Kaipa R, Danser ML. Efficacy of auditory-verbal therapy in children with hearing impairment: A systematic review from 1993 to 2015. Int J Pediatr Otorhinolaryngol. 2016 Jul;86:124-34. doi: 10.1016/j.ijporl.2016.04.033. Epub 2016 May 3. PMID 27260595
- [Background] Karpicke JD, Blunt JR, Smith MA. Retrieval-Based Learning: Positive Effects of Retrieval Practice in Elementary School Children. Front Psychol. 2016 Mar 11;7:350. doi: 10.3389/fpsyg.2016.00350. eCollection 2016. PMID 27014156
- [Background] Karpicke, J. D., Blunt, J. R., Smith, M. A., & Karpicke, S. S. (2014). Retrieval-based learning: The need for guided retrieval in elementary school children. Journal of Applied Research in Memory and Cognition, 3(3), 198-206.
- [Background] Knouse, L. E., Rawson, K. A., Vaughn, K. E., & Dunlosky, J. (2016). Does Testing Improve Learning for college students with attention-deficit/hyperactivity disorder? Clinical Psychological Science, 4(1), 136-143.
- [Background] Kyle FE, Harris M. Longitudinal patterns of emerging literacy in beginning deaf and hearing readers. J Deaf Stud Deaf Educ. 2011 Summer;16(3):289-304. doi: 10.1093/deafed/enq069. Epub 2011 Feb 9. PMID 21307357
- [Background] Leonard LB, Deevy P, Karpicke JD, Christ S, Weber C, Kueser JB, Haebig E. Adjective Learning in Young Typically Developing Children and Children With Developmental Language Disorder: A Retrieval-Based Approach. J Speech Lang Hear Res. 2019 Dec 5;62(12):4433-4449. doi: 10.1044/2019_JSLHR-L-19-0221. Print 2019 Dec 18. PMID 31805241
- [Background] Leonard LB, Karpicke J, Deevy P, Weber C, Christ S, Haebig E, Souto S, Kueser JB, Krok W. Retrieval-Based Word Learning in Young Typically Developing Children and Children With Developmental Language Disorder I: The Benefits of Repeated Retrieval. J Speech Lang Hear Res. 2019 Apr 15;62(4):932-943. doi: 10.1044/2018_JSLHR-L-18-0070. PMID 30986142
- [Background] Lipowski SL, Pyc MA, Dunlosky J, Rawson KA. Establishing and explaining the testing effect in free recall for young children. Dev Psychol. 2014 Apr;50(4):994-1000. doi: 10.1037/a0035202. Epub 2013 Dec 2. PMID 24294884
- [Background] Luckner JL, Cooke C. A summary of the vocabulary research with students who are deaf or hard of hearing. Am Ann Deaf. 2010 Spring;155(1):38-67. doi: 10.1353/aad.0.0129. PMID 20503907
- [Background] Lund E. Vocabulary Knowledge of Children With Cochlear Implants: A Meta-Analysis. J Deaf Stud Deaf Educ. 2016 Apr;21(2):107-21. doi: 10.1093/deafed/env060. Epub 2015 Dec 27. PMID 26712811
- [Background] Lund E, Miller C, Douglas WM, Werfel K. Teaching Vocabulary to Improve Print Knowledge in Preschool Children with Hearing Loss. Perspect ASHA Spec Interest Groups. 2020 Dec;5(6):1366-1379. doi: 10.1044/2020_persp-20-00023. Epub 2020 Aug 17. PMID 33981844
- [Background] Marsh EJ, Fazio LK, Goswick AE. Memorial consequences of testing school-aged children. Memory. 2012;20(8):899-906. doi: 10.1080/09658211.2012.708757. Epub 2012 Aug 15. PMID 22891857
- [Background] McDaniel J, Benitez-Barrera CR, Soares AC, Vargas A, Camarata S. Bilingual Versus Monolingual Vocabulary Instruction for Bilingual Children with Hearing Loss. J Deaf Stud Deaf Educ. 2019 Apr 1;24(2):142-160. doi: 10.1093/deafed/eny042. PMID 30597033
- [Background] McDaniel J, Camarata S, Yoder P. Comparing Auditory-Only and Audiovisual Word Learning for Children With Hearing Loss. J Deaf Stud Deaf Educ. 2018 Oct 1;23(4):382-398. doi: 10.1093/deafed/eny016. PMID 29767759
- [Background] McGregor KK, Gordon K, Eden N, Arbisi-Kelm T, Oleson J. Encoding Deficits Impede Word Learning and Memory in Adults With Developmental Language Disorders. J Speech Lang Hear Res. 2017 Oct 17;60(10):2891-2905. doi: 10.1044/2017_JSLHR-L-17-0031. PMID 28980007
- [Background] Nittrouer S, Lowenstein JH, Antonelli J. Parental Language Input to Children With Hearing Loss: Does It Matter in the End? J Speech Lang Hear Res. 2019 Dec 13;63(1):234-258. doi: 10.1044/2019_JSLHR-19-00123. Print 2020 Jan 22. PMID 31834998
- [Background] Qi S, Mitchell RE. Large-scale academic achievement testing of deaf and hard-of-hearing students: past, present, and future. J Deaf Stud Deaf Educ. 2012 Winter;17(1):1-18. doi: 10.1093/deafed/enr028. Epub 2011 Jun 28. PMID 21712463
- [Background] Reimer CK, Grantham H, Butler AC. The effect of retrieval practice on vocabulary learning for DHH children. J Deaf Stud Deaf Educ. 2024 Jun 24;29(3):377-387. doi: 10.1093/deafed/enae005. PMID 38330211
- [Background] Roberts MY. Parent-Implemented Communication Treatment for Infants and Toddlers With Hearing Loss: A Randomized Pilot Trial. J Speech Lang Hear Res. 2019 Jan 30;62(1):143-152. doi: 10.1044/2018_JSLHR-L-18-0079. PMID 30535174
- [Background] Ruben RJ. Language development in the pediatric cochlear implant patient. Laryngoscope Investig Otolaryngol. 2018 Apr 19;3(3):209-213. doi: 10.1002/lio2.156. eCollection 2018 Jun. PMID 30062136
- [Background] Werfel KL. Emergent Literacy Skills in Preschool Children With Hearing Loss Who Use Spoken Language: Initial Findings From the Early Language and Literacy Acquisition (ELLA) Study. Lang Speech Hear Serv Sch. 2017 Oct 5;48(4):249-259. doi: 10.1044/2017_LSHSS-17-0023. PMID 28973172
- [Background] Lehman M, Smith MA, Karpicke JD. Toward an episodic context account of retrieval-based learning: dissociating retrieval practice and elaboration. J Exp Psychol Learn Mem Cogn. 2014 Nov;40(6):1787-94. doi: 10.1037/xlm0000012. Epub 2014 May 5. PMID 24797442

DOCUMENTS (1):
  • Informed Consent Form (2025-02-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT05512000/ICF_000.pdf